CLINICAL TRIAL: NCT00878098
Title: Study of DDT and Loss of Clinically Recognized Pregnancies in South Africa
Brief Title: Study of DDT and Loss of Clinically-Recognized Pregnancies in South Africa
Status: Completed | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999909115; 09-E-N115
Record Dates: First submitted 2009-04-07; First posted 2009-04-08 (Estimated); Last update posted 2019-07-18 (Actual); Status verified 2019-07-12

CONDITIONS: Spontaneous Abortion; Malaria; Pregnancy Outcome; Stillbirth; HIV Infections
Keywords: DDT; Malaria; Pregnancy Outcome; Spontaneous Abortion; HIV; Pregnancy
MeSH Terms: conditions — Abortion, Spontaneous; Malaria; Stillbirth; HIV Infections

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Background:

* In some countries, such as South Africa, the pesticide DDT is an important chemical for control of malaria-carrying mosquitoes. However, there is little evidence about the effects that it might have on human health.
* DDT has been associated with miscarriage and fetal loss in areas with high levels of exposure, but more research is needed to determine what levels of exposure are associated with loss of pregnancies.

Objectives:

* To examine the relationship between pre-pregnancy levels of DDT in the blood and the loss of clinically recognized pregnancies.
* To conduct a pilot study to evaluate data collection procedures for future research.

Eligibility:

* Women between 20 and 30 years of age who are not currently pregnant and who reside in villages in the Vhembe District in the northeastern part of South Africa.

Design:

* Evaluation of eligibility:

  1. Short physical examination, with questionnaire about medical history, current living conditions, and daily life.
  2. Several blood samples will be taken for study and to test for anemia, elevated lead levels, malaria, syphilis, and human immunodeficiency virus (HIV).
* Half of the women will come from villages that are currently being sprayed with DDT, and half will come from villages that are not being sprayed.
* Evaluation before and during pregnancy for subjects who become pregnant:

  1. Blood and urine test, including urine pregnancy test.
  2. Questions about recent menstrual history and sexual activity.
  3. Questions about medical history, including treatment for malaria.
* Pregnancy follow-up study, including blood draws, will be conducted regardless of whether the pregnancy is carried to term.
* Researchers will assess and adjust study parameters as needed.

DETAILED DESCRIPTION:
In this study, the primary goal is to examine the relationship between DDT (dichlorodiphenyltrichloroethane) levels and the odds of loss of clinically-recognized pregnancies amongst women in Limpopo, South Africa. The initial protocol (which will be referred to as Part 1) planned to enroll 2,400 non-pregnant women, draw blood for measurement of DDT exposure, and follow 1,200 pregnant participants to ascertain occurrence of miscarriage. An initial two-year pilot of 850 non-pregnant women was proposed to evaluate field procedures, recruitment strategies and the reproducibility of DDT levels. Of the 444 women enrolled in the first 10 months of the pilot of Part 1, only 27 have become pregnant. Although the field procedures have been well executed, the number of pregnancies has been low. Based upon the experience to date, the approach taken so far is unlikely to generate enough pregnancies to monitor the occurrence of miscarriages. Therefore, the revised protocol (referred to as Part 2) will modify enrollment criteria to include only pregnant women who are in the early stages of pregnancy, confirmed by rising human chorionic gonadotropin (hCG) blood levels taken 1 week apart or pregnant women who have a pregnancy loss within 4 weeks of enrollment. Participants who were enrolled in Part 1 of the pilot, who are still not pregnant at implementation of Part 2 will be withdrawn from the study, while pregnant participants from Part 1 will continue to be followed. In Part 2, a total of 2,400 pregnant women will be enrolled. Only those who meet the follow-up criteria (n=1,200) will be followed to determine the outcome of pregnancy. The reproducibility study of DDT levels amongst a subset of 200 women will also be dropped and replaced with an analysis using specimens that were collected in Part 1.

ELIGIBILITY:
* ELIGIBILITY CRITERIA:

Enrollment criteria and follow-up criteria will be in two stages. Women will have to meet eligibility criteria to be enrolled for the study. Then, only those participants who meet the follow-up criteria will continue to be followed in the study until the end of their pregnancy. Those participants that do not meet the follow-up criteria will be withdrawn from the follow-up portion of the study.

ELIGIBILITY CRITERIA FOR ENROLLMENT

1. Aged 20-34 years
2. Plan to reside in the same (studied) village throughout participation in the study
3. Live in a village currently being studied
4. Have no previous pregnancy in the study
5. Have a positive spot pregnancy urine (hCG) test

ELIGIBILITY CRITERIA FOR FOLLOW-UP

1. Have two positive serum hCG tests at least one week apart, with the concentration of hCG in the second test being higher than that of the first, and who are still pregnant 4 weeks after the first blood test.
2. The first serum hCG test is positive and reports a pregnancy loss within the first 4 weeks after the first blood test. An Inexscreen urine pregnancy test confirms that the participant is no longer pregnant at the second clinic visit (1 week after the first blood test) or at the third clinic visit (4 weeks after the first blood test).

EXCLUSION CRITERIA FOR FOLLOW-UP

1. Have two positive serum hCG tests at least one week apart, with the concentration of hCG in the second test being equal or lower than that of the first, and are still pregnant 4 weeks after the first blood test.

Ages: 20 Years to 34 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 513 (Actual)
Dates: Start 2009-06-01; Study Completion 2019-07-12

CONTACTS AND LOCATIONS:
Overall Officials: Gitanjali Taneja, Ph.D., Principal Investigator — National Institute of Environmental Health Sciences (NIEHS)
Locations (1):
- Pretoria Academic Hospital, Thulamela Municipality, South Africa

REFERENCES:
- [Background] Aneck-Hahn NH, Schulenburg GW, Bornman MS, Farias P, de Jager C. Impaired semen quality associated with environmental DDT exposure in young men living in a malaria area in the Limpopo Province, South Africa. J Androl. 2007 May-Jun;28(3):423-34. doi: 10.2164/jandrol.106.001701. Epub 2006 Dec 27. PMID 17192596
- [Background] Cooper GS, Klebanoff MA, Promislow J, Brock JW, Longnecker MP. Polychlorinated biphenyls and menstrual cycle characteristics. Epidemiology. 2005 Mar;16(2):191-200. doi: 10.1097/01.ede.0000152913.12393.86. PMID 15703533
- [Background] Bouwman H, Cooppan RM, Becker PJ, Ngxongo S. Malaria control and levels of DDT in serum of two populations in Kwazulu. J Toxicol Environ Health. 1991 Jun;33(2):141-55. doi: 10.1080/15287399109531514. PMID 2051491